CLINICAL TRIAL: NCT06821178
Title: Stress, Memory, and Rumination in Maltreated Adolescents
Brief Title: My Life and My Experiences Project
Acronym: M&M Project
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Irvine (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Jodi Quas, Professor, University of California, Irvine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 4715; R01HD113752 (NIH)
Record Dates: First submitted 2025-02-06; First posted 2025-02-11 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-02

CONDITIONS: Stress and Memory in Adolescence

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- High Stress Condition (Experimental): High stress condition of Trier Social Stress Test - Modified
  Interventions: Behavioral: Acute stress manipulation
- Low Stress Condition (Experimental): Low stress condition of the Trier Social Stress Test-Modified
  Interventions: Behavioral: Acute stress manipulation

INTERVENTIONS:
Behavioral: Acute stress manipulation — Youth will be randomly assigned to the HS (high stress) or LS (low stress) TSST-M condition. The objective activities will be identical in the HS and LS conditions but the context will vary. The HS condition will be highly evaluative. The researcher will tell youth that they are being videotaped in order to code their behaviors later. The observers will maintain neutral expressions, provide instructions in a neutral tone, and avoid eye contact. In the LS condition, evaluative components are removed [31, 53]. Observers will be introduced as new, and the videotaping will be explained as a check to ensure that the observers follow instructions. The observers will appear disorganized while giving instructions, smile, and maintain an open body posture and eye contact.

SUMMARY:
Child maltreatment is one of the most formidable public health crises in the United States, affecting millions of youth each year. The adverse consequences of maltreatment for youth, as well as for their families and entire communities, are pervasive, costly, and enduring. To intervene and reduce these consequences, it is imperative that victims provide clear and accurate accounts of their prior experiences. Currently, considerable skepticism exists regarding maltreated youth's ability to provide such accounts, especially for experiences that were stressful, leading to youths' reports being challenged or not believed. It is possible that this skepticism is unwarranted, and maltreated youth actually demonstrate better memory than their non-maltreated counterparts, but only for stressful salient personal experiences. This project will ethically and rigorously test this possibility via a short-term longitudinal experimental investigation that compares the effects of acute stress on memory between maltreated and demographically matched non-maltreated 12-17-year-olds. In an initial in-person session, youth will be randomly assigned (equal maltreated and non-maltreated youth across age) to complete standardized salient personal activities that are experimentally manipulated to vary in whether they induce higher or lower levels of acute stress. Immediately afterward, youth will complete an encoding task comprised of positive, negative, and neutral images. In subsequent sessions (two remote and one in person) spanning approximately one month, youth's memory will be tested for the images via a recognition task asking them to discriminate previously seen from unseen images and for the personal activities via recall and direct questions that probe for the extent and accuracy of memory. Youth's rumination about the personal activities will also be measured. The project's main hypothesis is that maltreatment will lead to particularly robust memory for the personal activities, but only when the youth complete these under conditions of high stress. By contrast, because the emotional and neutral images are not personally meaningful, maltreatment is expected to constrain youth's memory performance for the images. It is also hypothesized that rumination will serve as an important mediator of the links between stress and memory for the higher stress personal activities, most notably in the maltreated youth. Overall, the project's results will provide much-needed knowledge about the precise ways that maltreatment shapes different facets of youth's memory, knowledge. This knowledge will be enormously valuable in improving trust in maltreated youth's reporting of stressful experiences and hence in directing interventions for victimized youth.

ELIGIBILITY:
Inclusion Criteria:

Ages 12-17 at start, half self reported or documented prior contact with social services/dependency court; half always lived with at least one biological parent

Exclusion Criteria:

Public speaking or math anxiety, cognitive impairments, head injuries, learning disabilities, steroid/hormonal treatments, or neuroendocrine diseases

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 400 (Estimated)
Dates: Start 2025-01-28 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Delarative recognition memory | 10 days from first session
  This memory measure reflects how well participants remember images that they encoded in Session 1. Participants are presented with previously seen and unseen images. Their job is to discriminate the two (i.e., say "old" for prior images and "new" for unseen images). Scores computed based on their responses include discriminability and response bias tendencies. These scores will be examined in relation to participants' maltreatment status and whether they encoded the images under high or low stress conditions.
Event Memory | 30 days from first session
  This memory measure reflects how well participants remember the entire first session, during which they had completed either the HS or LS TSST-M. Thus, of interest concerns differences in youth's memory for a stressful versus nonstressful prior salient experiences. Responses to recall and direct questions are coded for completeness and accuracy. These scores will be examined in relation to participants' maltreatment status and whether the original experience was higher versus lower stress.

SECONDARY OUTCOMES:
State Rumination | 10 days, 20 days, and 30 days from first session
  A measure of state rumination specifically about the first session, when participants completed the HS or LS TSST-M. Rumination is believed to operate as a mediator, influencing the relation between stress at encoding and later memory. Thus, preliminary analyses will evaluate whether youth who experienced the HS TSST-M ruminate more than youth who experienced the LS TSST-M, but also whether maltreated youth ruminate more than comparison youth.

CONTACTS AND LOCATIONS:
Locations (1):
- University of California, Irvine, Irvine, California, United States

IPD SHARING:
Plan to Share IPD: No